CLINICAL TRIAL: NCT04496752
Title: A Randomized Crossover Study to Assess the Reliability and Equivalence of Alternate Forms of the Digital Clock Drawing Test
Brief Title: Reliability and Equivalence of Alternate Forms of the Digital Clock Drawing Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linus Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: DCT216
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- DCTclock-pen first (Experimental): DCTclock-pen followed by DCTclock-tablet
  Interventions: Device: DCTclock
- DCTclock-tablet first (Experimental): DCTclock-tablet followed by DCTclock-pen
  Interventions: Device: DCTclock

INTERVENTIONS:
Device: DCTclock — Cognitive Test

SUMMARY:
Equivalence of DCTclock-pen and DCTclock-tablet will be tested in a randomized crossover trial.

DETAILED DESCRIPTION:
Randomized crossover trial consisting of two test visits separated by a washout period of 3 to 5 weeks. Subjects are randomized into two equal groups. Group 1 receives the digital pen (DCTclock-pen) version of the test at the first visit, with the tablet version (DCTclock-tablet) given at the second visit; Group 2 receives DCTclock-tablet at the first visit, followed by DCTclock-pen at the second visit. At Visit 1 (day 0), eligibility is assessed and a version of the DCTclock test is administered based on the group allocation. A battery of Linus Platform tests and reference standard tests are also administered. At visit 2 (day 21-35), eligibility is assessed and the alternate version of the DCTclock test is administered based on the group allocation. A battery of Linus Platform tests is also administered, together with reference standard tests. Equivalence of DCTclock-pen and DCTclock-tablet will be tested. Linus Platform test data will also be collected to develop novel measures of cognitive and motor function and assess their accuracy in detecting impairment, construct validity, and test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

* 55-95 years old

Exclusion Criteria:

* Ineligible for written informed consent
* Impairment of the writing hand that precludes ability to perform the study tasks
* Impaired manual dexterity in the writing hand
* Impaired vision in both eyes
* Under the influence of recreational drugs or alcohol at the time of the visit.
* Current or recent participation in a clinical trial that includes the use of a drug or intervention to alter cognitive function.
* Recent (within the last 6 months) cognitive testing with a Clock Drawing Test.
* Visit 2 Only- Self-reported change (addition or discontinuation) of the following medications between visit 1 and visit 2; Timolol (eye drop), Benadryl, beta blockers, steroids or over the counter medications for sleep (PM varieties).

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Pascual-Leone, MD, Study Chair — Linus Health
Locations (2):
- United States (2):
  - Clincloud Research, Maitland, Florida
  - Clinilabs, Eatontown, New Jersey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by referral from neurology clinics at 2 study sites. The first participant was enrolled in December 2020, and the last participant was enrolled in May 2021.
Pre-assignment Details: Screening for inclusion criteria was conducted at the first study session after enrollment and prior to randomization. Of 200 enrolled participants, 195 met inclusion criteria and were randomized to groups.
Period: First Assessment
Arm/Group | DCTclock-pen First | DCTclock-tablet First
Started | 97 | 98
Completed | 97 | 98
Not Completed | 0 | 0
Period: Second Assessment
Arm/Group | DCTclock-pen First | DCTclock-tablet First
Started | 97 | 98
Second Visit Begun | 92 | 95
Completed | 92 | 95
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 3 | 3
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DCTclock-pen First | DCTclock-tablet First | Total
Number analyzed (Participants) | 97 | 98 | 195
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 58 | 110
  >=65 years | 45 | 40 | 85
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 62 | 118
  Male | 41 | 36 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 19 | 38
  Not Hispanic or Latino | 78 | 79 | 157
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 24 | 47
  White | 69 | 71 | 140
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Handedness [Count of Participants; unit: Participants]
  Left | 9 | 10 | 19
  Right | 88 | 87 | 175
  Ambidextrous | 0 | 1 | 1
Education [Count of Participants; unit: Participants]
  Less than High School | 6 | 6 | 12
  High School Degree | 16 | 24 | 40
  Some College | 35 | 30 | 65
  College Degree or Higher | 40 | 38 | 78
Dementia Medication Usage [Count of Participants; unit: Participants]
  Aricept (Donepezil): Currently | 4 | 4 | 8
  Aricept (Donepezil): Previously | 2 | 1 | 3
  Aricept (Donepezil): Never | 91 | 93 | 184
  Namenda (Mematine): Currently | 5 | 2 | 7
  Namenda (Mematine): Previously | 0 | 1 | 1
  Namenda (Mematine): Never | 92 | 95 | 187
  Axona: Currently | 0 | 0 | 0
  Axona: Previously | 0 | 0 | 0
  Axona: Never | 97 | 98 | 195
  Exelon (Rivastigmine): Currently | 2 | 0 | 2
  Exelon (Rivastigmine): Previously | 0 | 0 | 0
  Exelon (Rivastigmine): Never | 95 | 98 | 193
  Razadyne (Galantamine): Currently | 0 | 0 | 0
  Razadyne (Galantamine): Previously | 0 | 0 | 0
  Razadyne (Galantamine): Never | 97 | 98 | 195
Mini-Mental State Exam (MMSE) Score [Mean (Standard Deviation); unit: units on a scale] — The Mini-Mental State Examination (MMSE) Score is an assessment of cognitive impairment, consisting of a standardized set of tasks. MMSE scores range 0-30, with lower scores indicating greater impairment. The total score is the sum of subscales (ranges in parentheses): Orientation to Time (0-5), Orientation to Place (0-5), Registration (0-3), Attention and Calculation (0-5), Recall (0-3), Naming (0-2), Repetition (0-1), Comprehension (0-3), Reading (0-1), Writing (0-1), Drawing (0-1).
  units on a scale
    Orientation to Time | 4.8 (0.5) | 4.7 (0.8) | 4.7 (0.7)
    Orientation to Place | 4.4 (0.7) | 4.3 (0.8) | 4.4 (0.7)
    Registration | 3.0 (0.0) | 3.0 (0.1) | 3.0 (0.1)
    Attention and Calculation (WORLD) | 4.6 (0.9) | 4.7 (0.7) | 4.7 (0.8)
    Recall | 2.6 (0.7) | 2.7 (0.7) | 2.6 (0.7)
    Naming | 2.0 (0.1) | 2.0 (0.0) | 2.0 (0.1)
    Repetition | 0.8 (0.4) | 0.8 (0.4) | 0.8 (0.4)
    Comprehension | 3.0 (0.1) | 2.9 (0.3) | 3.0 (0.2)
    Reading | 1.0 (0.1) | 1.0 (0.0) | 1.0 (0.1)
    Writing | 1.0 (0.1) | 1.0 (0.1) | 1.0 (0.1)
    Drawing | 0.8 (0.4) | 0.8 (0.4) | 0.8 (0.4)
    Total | 27.9 (2.2) | 27.9 (2.4) | 27.9 (2.3)
Hamilton-Veale Contrast Sensitivity Score [Mean (Standard Deviation); unit: units on a scale] — The Hamilton-Veale Contrast Sensitivity Score is an assessment of visual sensitivity to contrast. It is measured with a standardized chart presenting a grid of letters with varying contrast relative to a white background. It is assessed separately for the left and right eyes, and for both eyes together (binocular). Scores range 0-16, with a higher score indicating greater sensitivity and an ability to detect lower contrast.
  units on a scale
    Left | 10.6 (1.8) | 10.7 (2.4) | 10.7 (2.1)
    Right | 10.6 (1.7) | 10.6 (2.5) | 10.6 (2.1)
    Binocular | 11.4 (1.1) | 11.6 (1.1) | 11.5 (1.1)
Purdue Pegboard Score [Mean (Standard Deviation); unit: units on a scale] — The Purdue Pegboard Test is an assessment of manual dexterity and motor coordination. The score (ranging 0-25) is the number of pegs a subject is able to place in a grooved board within a time limit. A higher score (more pegs) indicates greater dexterity. The assessment is performed separately for each hand, and for both hands together.
  units on a scale
    Left | 10.3 (2.1) | 10.4 (2.2) | 10.4 (2.1)
    Right | 11.0 (2.4) | 11.3 (2.5) | 11.1 (2.5)
    Both Hands | 10.7 (5.0) | 11.7 (5.2) | 11.2 (5.1)
Medical History [Count of Participants; unit: Participants] — # of participants reporting history of relevant conditions
  Participants
    Parkinson's Disease and Related Conditions: Currently | 1 | 0 | 1
    Parkinson's Disease and Related Conditions: Previously | 0 | 0 | 0
    Parkinson's Disease and Related Conditions: Never | 96 | 98 | 194
    Sleep Apnea: Currently | 9 | 16 | 25
    Sleep Apnea: Previously | 1 | 2 | 3
    Sleep Apnea: Never | 87 | 80 | 167
    Stroke or TIA: Currently | 1 | 0 | 1
    Stroke or TIA: Previously | 5 | 5 | 10
    Stroke or TIA: Never | 91 | 93 | 184
    Liver or Kidney Disease: Currently | 5 | 2 | 7
    Liver or Kidney Disease: Previously | 0 | 1 | 1
    Liver or Kidney Disease: Never | 92 | 95 | 187
    Tremor: Currently | 1 | 1 | 2
    Tremor: Previously | 1 | 1 | 2
    Tremor: Never | 95 | 96 | 191
    Brain Tumor: Currently | 0 | 1 | 1
    Brain Tumor: Previously | 1 | 0 | 1
    Brain Tumor: Never | 96 | 97 | 193
    Psychiatric Disorder (including Anxiety/Depression): Currently | 14 | 20 | 34
    Psychiatric Disorder (including Anxiety/Depression): Previously | 4 | 3 | 7
    Psychiatric Disorder (including Anxiety/Depression): Never | 79 | 75 | 154
    Dementia (any type): Currently | 3 | 1 | 4
    Dementia (any type): Previously | 0 | 1 | 1
    Dementia (any type): Never | 94 | 96 | 190
    Diabetes: Currently | 32 | 28 | 60
    Diabetes: Previously | 1 | 0 | 1
    Diabetes: Never | 64 | 70 | 134
    Mild Cognitive Impairment (MCI): Currently | 0 | 2 | 2
    Mild Cognitive Impairment (MCI): Previously | 0 | 0 | 0
    Mild Cognitive Impairment (MCI): Never | 97 | 96 | 193
    Traumatic brain injury (with loss of consciousness): Currently | 0 | 1 | 1
    Traumatic brain injury (with loss of consciousness): Previously | 5 | 4 | 9
    Traumatic brain injury (with loss of consciousness): Never | 92 | 93 | 185

OUTCOME MEASURES:

1. Primary Outcome: Equivalence of DCTclock-pen and DCTclock-tablet in Assessing Cognitive Impairment
Description: Equivalence of DCTclock-pen and DCTclock-tablet in assessing cognitive impairment, as measured by comparison of agreement with MMSE.
Time Frame: 5 weeks
Population: Analysis includes only assessments from participants who: (1) completed both assessment sessions; and (2) produced clocks from both assessments which could be analyzed to give a valid score. Of participants who completed both sessions, 170 of 187 produced two analyzable clocks and were included in analysis (84 of 92 in the pen-first group, and 86 of 95 in the tablet-first group).
Measure: Number (90% Confidence Interval); unit: Cohen's Kappa Coefficient
Units Other Than Participants: Assessments
Groups:
- DCTClock-pen: Assessments with the DCTClock-pen format, from participants who completed assessments with both DCTClock-pen and DCTClock-tablet.
  Assessments from participants who failed to complete either of the formats, due to protocol deviations and/or technical failure, were excluded.
- DCTClock-tablet: Assessments with the DCTClock-tablet format, from participants who completed assessments with both DCTClock-pen and DCTClock-tablet.
  Assessments from participants who failed to complete either of the formats, due to protocol deviations and/or technical failure, were excluded.
Arm/Group | DCTClock-pen | DCTClock-tablet
Number analyzed (Participants) | 170 | 170
Number analyzed (Assessments) | 170 | 170
Cohen's Kappa Coefficient | 0.16 [0.05 to 0.27] | 0.23 [0.12 to 0.33]
Statistical Analysis 1: Comparison: DCTClock-pen vs DCTClock-tablet; Test type: Equivalence — Weighted Cohen's kappa statistics were computed between DCTClock-pen and MMSE, and between DCTClock-tablet and MMSE. A TOST (two one-sided test) of equivalence was planned, with a difference in kappa of 0.2 specified a priori as significant; Difference in Cohen's Kappa = 0.07, 90% CI 2-sided [-0.05 to 0.19] — The difference is Cohen's kappa is (tablet - pen). The confidence interval is estimated with a nonparametric bootstrap (5000 samples)

2. Secondary Outcome: Number of Participants With Device-Related and Non-Device Related Adverse Events
Description: Number of serious device-related adverse events. See adverse events section for full reporting of adverse events, including both device-related and non-device related.
Time Frame: 5 weeks
Population: All participants who passed screening and were enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | DCTclock-pen First | DCTclock-tablet First
Number analyzed (Participants) | 97 | 98
Participants
  During Visit 1: Device-Related Adverse Event | 0 | 0
  During Visit 1: Other Adverse Event | 0 | 0
  During Visit 1: No Adverse Event | 97 | 98
  Between Visits: Device-Related Adverse Event | 0 | 0
  Between Visits: Other Adverse Event | 7 | 1
  Between Visits: No Adverse Event | 90 | 97
  During Visit 2: Device-Related Adverse Event | 0 | 0
  During Visit 2: Other Adverse Event | 0 | 1
  During Visit 2: No Adverse Event | 97 | 97
  Overall: Device-Related Adverse Event | 0 | 0
  Overall: Other Adverse Event | 7 | 2
  Overall: No Adverse Event | 90 | 96

3. Primary Outcome: Equivalence of DCTclock-pen and DCTclock-tablet in Assessing Cognitive Impairment (Correlation)
Description: Equivalence of DCTclock-pen and DCTclock-tablet in assessing cognitive impairment, as measured by comparison of correlation with MMSE.
Time Frame: 5 weeks
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: correlation coefficient
Units Other Than Participants: Assessments
Arm/Group | DCTClock-pen | DCTClock-tablet
Number analyzed (Participants) | 170 | 170
Number analyzed (Assessments) | 170 | 170
correlation coefficient
  Pearson Correlation | 0.31 [0.17 to 0.43] | 0.37 [0.25 to 0.49]
  Spearman Correlation | 0.29 [0.17 to 0.41] | 0.36 [0.24 to 0.46]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the start of the first study visit to the end of the second and last visit (3-5 weeks subsequent).
Description: Investigators completed a case report form (CRF), including a structured adverse event report, at each study visit.
Groups:
- DCTclock-pen First, DCTclock-pen Visit: The DCTclock-pen visit for participants who were assessed with the DCTclock-pen in the first visit, and DCTclock-tablet in the second visit (i.e., Visit 1).
- DCTclock-tablet First, DCTclock-tablet Visit: The DCTclock-tablet visit for participants who were assessed with the DCTclock-tablet in the first visit, and DCTclock-pen in the second visit (i.e., Visit 1).
- DCTclock-pen First, DCTclock-tablet Visit: The DCTclock-tablet visit for participants who were assessed with the DCTclock-pen at the first visit, and the DCTclock-tablet second visit (i.e., Visit 2).
- DCTclock-tablet First, DCTclock-pen Visit: The DCTclock-pen visit for participants who were assessed with the DCTclock-tablet at the first visit, and the DCTclock-pen at the second visit (i.e., Visit 2).
- DCTclock-pen First, Between Visits: Captures any reported events that occurred between the two study visits, for participants who were assessed with the DCTclock-pen at the first visit, and the DCTclock-tablet at the second visit.
- DCTclock-tablet First, Between Visits: Captures any reported events that occurred between the two study visits, for participants who were assessed with the DCTclock-tablet at the first visit, and the DCTclock-pen at the second visit.
Arm/Group | DCTclock-pen First, DCTclock-pen Visit | DCTclock-tablet First, DCTclock-tablet Visit | DCTclock-pen First, DCTclock-tablet Visit | DCTclock-tablet First, DCTclock-pen Visit | DCTclock-pen First, Between Visits | DCTclock-tablet First, Between Visits
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/98 | 0/97 | 0/98 | 1/97 | 0/98
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/98 | 0/97 | 0/98 | 3/97 | 0/98
Other Adverse Events (participants affected / at risk) | 0/97 | 0/98 | 0/97 | 1/98 | 4/97 | 1/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DCTclock-pen First, DCTclock-pen Visit (N=97) | DCTclock-tablet First, DCTclock-tablet Visit (N=98) | DCTclock-pen First, DCTclock-tablet Visit (N=97) | DCTclock-tablet First, DCTclock-pen Visit (N=98) | DCTclock-pen First, Between Visits (N=97) | DCTclock-tablet First, Between Visits (N=98)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA — Unknown cause; details not provided by next of kin; incident occurred between visits and was unrelated to study procedures
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA — Reported as "shortness of breath"
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DCTclock-pen First, DCTclock-pen Visit (N=97) | DCTclock-tablet First, DCTclock-tablet Visit (N=98) | DCTclock-pen First, DCTclock-tablet Visit (N=97) | DCTclock-tablet First, DCTclock-pen Visit (N=98) | DCTclock-pen First, Between Visits (N=97) | DCTclock-tablet First, Between Visits (N=98)
Eye infection (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — worsening of existing condition
Covid Vaccine Side Effects (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — self-reported, detail not specified
Vertigo (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Reported as "dizziness"
Fracture of Bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT04496752/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT04496752/SAP_001.pdf